CLINICAL TRIAL: NCT05748080
Title: Two Apples a Day, Keep the Doctor Away?
Brief Title: The Apple Study: Two Apples a Day, Keep the Doctor Away?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: METC22-064
Record Dates: First submitted 2023-01-30; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Microbial Colonization; Enzyme Overdose
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apple intervention (Experimental): the eating of 2 apples a day for a period of 6 weeks
  Interventions: Other: Eating apples

INTERVENTIONS:
Other: Eating apples — the eating of 2 apples a day for a period of 6 weeks

SUMMARY:
The goal of this clinical trial is to learn about the gut microbiome in healthy postmenopausal women aged 50-64. The main questions it aims to answer are:

* Investigate whether the activity of the bacterial enzyme β-glucuronidase and the abundance of β-glucuronidase-producing bacteria could be decreased by ingestion of 2 apples a day for a period of 6 weeks
* Examine changes in gut microbiota composition, diversity, and functional capacity
* Examine feasibility of eating 2 apples a day for a period of 6 weeks

Participants will eat 2 apples a day for a period of 6 weeks.

Six weeks includes the period from the start of the study and gathering of baseline characteristics/questionnaires till the finish.

DETAILED DESCRIPTION:
It is know that estrogen levels decrease after menopause. There are many different factors affecting these levels though; the gut microbiome has been identified as one of these. Not only the composition of the gut microbiota plays a role here, but also its activity is of special interest. The gut microbiota for instance produces the bacterial enzyme β-glucuronidase which has been shown to de-conjugate biliary excreted estrogens, leading to reactivation and reabsorption of estrogens into the bloodstream. It might be expected that this reabsorption results in elevated blood estrogen levels. Elevated levels of estrogen have been linked to not only development but also recurrence of breast cancer.

Apples are known for their pectin which has prebiotic properties and a potential decreasing effect on β-glucuronidase activity. In vitro studies and animal studies have already shown the β-glucuronidase decreasing impact of pectin. In humans this was never examined before.

This study aims to investigate whether it is possible to lower the activity of the bacterial enzyme β-glucuronidase and the abundance of β-glucuronidase-producing bacteria by a simple dietary intervention. This dietary intervention consists of the ingestion of two whole apples a day, one in the morning and one in the evening, during the period of 6 weeks. Thereby this study aims to examine the feasibility of this intervention.

It is hypothesized that

1. this is a feasible intervention
2. this results in a decrease in the activity of the bacterial enzyme β-glucuronidase and the abundance of β-glucuronidase-producing bacteria. Which would be in line with the findings of in vitro and animal studies and
3. an increase in microbial diversity

ELIGIBILITY:
Inclusion Criteria:

* Age 50-64
* Postmenopausal women
* Recent negative breast cancer screening (< 6 months)

Exclusion Criteria:

* The regular consumption of one ore more apples a day
* Previous gastrointestinal surgery (excl. appendix surgery)
* Any type of cancer in history, except for basal cell carcinoma (BCC)
* Inflammatory bowel disease
* Mammography older than 6 months
* Antibiotic use within three months before fecal sampling
* Physically or mentally incapable or incompetent to sign informed consent
* Known apple allergy or complaints matching with apple allergy
* Less good dental state

Ages: 50 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
The activity of the bacterial enzyme β-glucuronidase and the abundance of β-glucuronidase-producing bacteria | 6 weeks per patient
  This will be measured in fecal samples by using a validated β-glucuronidase enzyme activity assay, which is based on previous studies.
Changes in gut microbiota composition, diversity, and functional capacity | 6 weeks per patient
  Gut microbiota composition, diversity
Feasibility of eating 2 apples a day for a period of 6 weeks | 6 weeks per patient
  feasibility

SECONDARY OUTCOMES:
Fecal levels of short-chain fatty acids (SCFA) | 6 weeks per patient
  SCFA
Dietary intake, medication, stool classification and frequency, blood pressure, weight, length and quality of life before and after the intervention | 6 weeks per patient
  diet/medication etc

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein Smidt, prof. dr., Principal Investigator — Maastricht University Medical Center